CLINICAL TRIAL: NCT00664391
Title: Monocentric Study, Phase III, for Safety Dermatological Evaluation: Acceptability With Gynecological Follow up - Dermacyd Breeze
Brief Title: Safety Dermatological Evaluation: Acceptability With Gynecological Follow up - Dermacyd Breeze
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: GMA-CO/Medical Director, sanofi-aventis administrative office France
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LACAC_L_03746
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2009-02-10 (Estimated); Status verified 2009-02

CONDITIONS: Hygiene
MeSH Terms: interventions — Lactic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Lactic acid (Dermacid)

INTERVENTIONS:
Drug: Lactic acid (Dermacid) — Liquid soup to be applied in the external genital area, in small quantity, with abundantly rinse after use, during 21 days

SUMMARY:
The purpose of this study is to demonstrate the safety of the gynecological formulation in normal and usual usage condition of Dermacyd Breeze.

ELIGIBILITY:
Inclusion Criteria:

* Integral skin test in the region;

Exclusion Criteria:

* Lactation or gestational risk or gestation;
* Use of Anti-inflammatory or immunosuppression drugs 1 month before the study;
* Topical medication use at the region to be treated;
* Cutaneous disease or active gynecological disease which may interfere in study results;
* Personal history of allergic disease at the area to be treated;
* Allergic or atopic history;

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-01; Primary Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Adverse events and their intensity and their association with the treatment. | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, Study Director — Sanofi-aventis administrative office Brazil
Locations (1):
- Sanofi-aventis, São Paulo, São Paulo, Brazil